CLINICAL TRIAL: NCT02682277
Title: Efficacy of Polyglucosamine for Weight Loss - in a Randomized, Double-blind, Placebo-controlled Clinical Investigation
Brief Title: Efficacy of Polyglucosamine Long Term Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Certmedica International GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 003/14; U111111292405 (Other: WHO)
Record Dates: First submitted 2016-02-10; First posted 2016-02-15 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-02

CONDITIONS: Obesity
Keywords: obesity; body weight; overweight; weight loss; polyglucosamine; L112; caloric restriction; physical activity
MeSH Terms: conditions — Obesity; Body Weight; Overweight; Weight Loss; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical device polyglucosamine (Active Comparator): 2 times daily 2 polyglucosamine tablets with the two main meals with 10 % reduction of caloric intake with no increase of physical activity
  Interventions: Device: polygucosamine
- Placebo (Placebo Comparator): 2 times daily 2 placebo tablets with the two main meals with 10 % reduction of caloric intake with no increase of physical activity
  Interventions: Other: placebo

INTERVENTIONS:
Device: polygucosamine — 2 times daily 2 polyglucosamine tablets with the two main meals with 10 % reduction of caloric intake with no increase of physical activity.
  Other Names: ß-1,4 polymer of D-glucosamine and N-acetyl-D-glucosamine
  Arms: Medical device polyglucosamine
Other: placebo — 2 times daily 2 placebo tablets with the two main meals with 10 % reduction of caloric intake with no increase of physical activity.
  Arms: Placebo

SUMMARY:
The polyglucosamine, specification L112, is a medical device and in this clinical trial used for weight reduction in moderately obese participants following a long term treatment lasting 12 months. The rationale for this study is to show that overweight can be reduced by taking 2 times daily 2 tablets with the main meals.

DETAILED DESCRIPTION:
Two groups of subjects were compared. A comparable diet condition, consisting of 10 % reduction of caloric intake was followed, according to a questionnaire based on the weekly number of servings. No modification of physical activity was requested.

One group had to take the polyglucosamine tablets and the other group placebo tablets for at least 12 months. It is known, that polyglucosamine is a fat binder acting in a physical-chemical manner, the positive charged fiber is bound to the negative charged dietary fat and this complex is unable to pass the gut wall into the body but is naturally excreted,hence this energy is not available. Therefore, this medical device should show a measurable reduction in body weight.

ELIGIBILITY:
Inclusion Criteria:

* BMI >30 and < 35
* waist circumference of more than 88 cm for women and greater than 102 for men

Exclusion Criteria:

* pregnancy or breast-feeding
* alcohol abuse
* drug abuse or drug addiction
* inability to fulfill the criteria of the trial protocol
* cancer diseases
* malignant tumors
* pre-existence of chronic intestinal disease
* known hypersensitivity reactions to crustaceans

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who could reduce their body weight by 10 or more per cent compared to the initial body weight. | 12 months

SECONDARY OUTCOMES:
Change of body weight in kg | 12 months
Change of BMI | 12 monts
Reduction of waist circumference | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gianni Belcaro, Principal Investigator — Irwine Labs University of Chieti; Umberto Cornelli, MD, Study Director — Loyola University School of Medicine-Chicago
Locations (1):
- MAP Center, Rende, Cosenza, Italy

IPD SHARING:
Plan to Share IPD: No